CLINICAL TRIAL: NCT05145309
Title: Value of Potassium Magnesium Citrate in Preventing and Treating Hypertension in African Americans
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Wanpen Vongpatanasin, Professor of Medicine, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: STU-2021-0912
Record Dates: First submitted 2021-11-10; First posted 2021-12-06 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — potassium-magnesium citrate

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The study supplement will be dispensed in a blinded manner.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Potassium Magnesium Citrate (KMgCit) first then Placebo (Experimental): Patients will be asked to take KMgCit ( Sterling Pharmaceutical Services) first for 4 weeks. The content of each sachet will be dissolved in 250 ml water and will be drunk with breakfast and again with dinner during the KMgCit Phase, to deliver 40 meq K, 20 meq Mg and 74 meq citrate per day. Then, subjects will be asked to take Placebo packaged in an identical sachet by dissolving in 250 ml water and drink it with breakfast and again with dinner for 4 weeks
  Interventions: Drug: KMgCit; Drug: Placebo
- Placebo first then KMgCit (Experimental): Patients will be asked to take Placebo packaged in an identical sachet by dissolving in 250 ml water and drink it with breakfast and again with dinner for 4 weeks. Then, subjects will be asked to take KMgCit (Sterling Pharmaceutical Services, Dupo, IL) after dissolving in 250 ml water and drink it with breakfast and again with dinner for 4 weeks
  Interventions: Drug: KMgCit; Drug: Placebo

INTERVENTIONS:
Drug: KMgCit — Supplement that provide K, Mg, and citrate
  Other Names: Potassium Magnesium Citrate
Drug: Placebo — Power with identical appearance to KMgCit

SUMMARY:
In the DASH (Dietary Approaches to Stop Hypertension) trials, a diet rich in fruits, vegetables, nuts and dairy products, and limited in fat content, was shown to be useful in controlling hypertension, particularly in African Americans (AA). Key components of such a diet are potassium, magnesium, and alkali, each of which has been implicated in lowering blood pressure. In the original IND 116,208, the investigators explored whether potassium-magnesium citrate (KMgCit) as a powder pharmaceutical formulation (dissolved in water before ingestion) could serve as a surrogate for the DASH diet and would lower blood pressure among patients with pre- or Stage I hypertension. Unfortunately, previous studies did not include adequate number of African American patients.

DETAILED DESCRIPTION:
This is a double blind, randomized crossover trial comprising two phases: Placebo Phase (microcrystalline cellulose in water) and KMgCit Phase (KMgCit powder in water) to investigate the use of KMgCit in lowering blood pressure and reducing arterial stiffness. One half of the subjects will undergo the Placebo phase first followed by the KMgCit phase. The other half will undergo the KMgCit phase first followed by the Placebo phase. Each phase is 4 weeks in duration with at least 1 week washout between phases.

Forty-five African American patients of either sex with pre- or Stage I hypertension, with systolic blood pressure of 120-139 mm or diastolic of < 90 mmHg according the 2017 ACC/AHA high BP guideline, will be recruited into the trial, with the expectation that 36 patients would complete both phases of the trial (assuming 20% dropout). They may be AA adult men or women (> 21 years of age). They may be on ACE inhibitor or ARB, but not on spironolactone or diuretic. Excluded will be patients with diabetes mellitus, renal impairment, heart disease, chronic NSAID use, gastrointestinal reflux disease requiring treatment with acid reducing agent of antacid more than once a week, esophageal-gastric ulcer, chronic diarrhea, hyperkalemia, abnormal liver function test, subjects who require potassium supplementation on a regular basis for any reason, pregnancy, history of major depression, bipolar disorder or schizophrenia, and history of substance abuse

ELIGIBILITY:
Inclusion Criteria:

-African American patients with pre- or Stage I hypertension, with systolic blood pressure of 120-139 mm or diastolic BP of < 90 mmHg.

Exclusion Criteria:

* Diabetes mellitus,
* Renal impairment (serum creatinine > 1.4 mg/dL),
* Any heart diseases such as congestive heart failure or sustained arrhythmia,
* Chronic NSAID use,
* Treatment with diuretics, including spironolactone
* Gastroesophageal reflux disease (GERD) requiring treatment with acid reducing agent or antacid more than once a week,
* Esophageal-gastric ulcer,
* Chronic diarrhea,
* Hyperkalemia (serum K > 5.0 mmol/L),
* Abnormal liver function test (AST or ALT above upper limit of normal range),
* Subjects who require any potassium supplement on a regular basis for any reason,
* Pregnancy,
* History of major depression, bipolar disorder, or schizophrenia, and
* History of substance abuse.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2026-11-15 (Estimated); Primary Completion 2031-12-01 (Estimated); Study Completion 2032-12-01 (Estimated)

PRIMARY OUTCOMES:
24-hour systolic blood pressure (24h SBP) | 4 weeks
  24-hour blood pressures will be recorded using the Spacelab ambulatory oscillometric blood pressure monitor (ABPM) (Spacelabs Medical, Issaquah, WA). Recordings will be made every 20 minutes during the day and every 30 minutes at night. Average data will be calculated for each patient and reported as mmHg.

SECONDARY OUTCOMES:
central systolic blood pressure (cSBP) | 4 weeks
  Arterial tonometry and simultaneous ECG will be obtained from the brachial, radial, femoral and carotid arteries noninvasively on the skin using a custom pulse transducer device manufactured by Cardiovascular Engineering, Inc. Carotid systolic BP will be used as central systolic blood pressure. The body surface distances from the suprasternal notch to the brachial (SSN-B), radial (SSN-R), femoral (SSN-F) to calculate carotid to femoral pulse wave velocity. Data will be reported as mmHg.
pulse wave velocity | 4 weeks
  Arterial tonometry and simultaneous ECG will be obtained from the brachial, radial, femoral and carotid arteries noninvasively on the skin, using a custom pulse transducer device manufactured by Cardiovascular Engineering, Inc. Carotid systolic BP will be used as central systolic blood pressure. The body surface distances from the suprasternal notch to the brachial (SSN-B), radial (SSN-R), femoral (SSN-F) to calculate carotid to femoral pulse wave velocity. Data will be reported as meter/second.
augmentation index | 4 weeks
  Arterial tonometry and simultaneous ECG will be obtained from the brachial, radial, femoral and carotid arteries noninvasively on the skin, using a custom pulse transducer device manufactured by Cardiovascular Engineering, Inc. Carotid systolic BP will be used as central systolic blood pressure. The computer program will analyze carotid waveform to calculate augmentation index. data will be reported as %.
FGF23 | 4 weeks
  Blood samples will be obtained after 4 weeks of study intervention for measurement of FGF23 concentration, a hormone involved in bone metabolism
klotho | 4 weeks
  Blood samples will be obtained after 4 weeks of study intervention for measurement of klotho concentration, a hormone involved in bone metabolism

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-15): https://cdn.clinicaltrials.gov/large-docs/09/NCT05145309/Prot_SAP_000.pdf